CLINICAL TRIAL: NCT06605144
Title: Canadian Critical Care Comparative Effectiveness Platform(e) d'Évaluation Clinique Comparée en Soins Critiques (CEPEC)
Brief Title: Canadian Critical Care Comparative Effectiveness Platform
Acronym: CEPEC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-31-2025-5600
Record Dates: First submitted 2024-09-10; First posted 2024-09-20 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Intensive Care Unit ICU; Vasopressor; Platelet
Keywords: ICU; Adaptive platform trial; Vasopressor; Platelet

STUDY DESIGN:
Intervention Model Description: Adaptive Bayesian Platform trial evaluating multiple interventions in multiple domains.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vasopressor (Other): Participants will receive vasopressor(s) and their mean arterial pressure will be titrated according to the group they are randomized to (group 1: 56-60 mmHg; group 2: 61-65 mmHg; group 3: 66-70 mmHg; group 4: 71-75 mmHg). Physicians will have the liberty of restricting the randomization to at least 2 contiguous ranges
  Interventions: Drug: 1- Vasopressor - Mean arterial pressure 56-60; Drug: 2- Vasopressor - Mean arterial pressure 61-65; Drug: 3- Vasopressor - Mean arterial pressure 66-70; Drug: 4- Vasopressor - Mean arterial pressure 71-75
- Platelet (Other): Thrombocytopenic intensive care unit (ICU) patients (platelet count <50×109/L) with a planned low-moderate bleeding-risk procedure will be randomized to one of five equally spaced platelet thresholds (less than 10 x 109/L, less than 20 x 109/L, less than 30 x 109/L, less than 40 x 109/L, less than 50 X 109/L) below which they will receive prophylactic platelet transfusions before any low-moderate bleeding-risk procedure occurring during the ICU episode up to ICU day 90. Once randomized, the clinical team will administer a platelet transfusion according to the assigned threshold and the most recent platelet count at the time of the planned procedure.
  Interventions: Other: 1- Platelet less than 10 x 109/L; Other: 2- Platelet less than 20 x 109/L; Other: 3- Platelet less than 30 x 109/L; Other: 4- Platelet less than 40 x 109/L; Other: 5- Platelet less than 50 x 109/L

INTERVENTIONS:
Drug: 1- Vasopressor - Mean arterial pressure 56-60 — Vasopressor(s) will be titrated according to 56-60 range.
  Arms: Vasopressor
Drug: 2- Vasopressor - Mean arterial pressure 61-65 — Vasopressor(s) will be titrated according to 61-65 range.
  Arms: Vasopressor
Drug: 3- Vasopressor - Mean arterial pressure 66-70 — Vasopressor(s) will be titrated according to 66-70 range.
  Arms: Vasopressor
Drug: 4- Vasopressor - Mean arterial pressure 71-75 — Vasopressor(s) will be titrated according to 71-75 range.
  Arms: Vasopressor
Other: 1- Platelet less than 10 x 109/L — Once randomized, the participant will receive a platelet transfusion if their most recent platelet count is less than 10 x 109/L at the time of the planned procedure.
  Arms: Platelet
Other: 2- Platelet less than 20 x 109/L — Once randomized, the participant will receive a platelet transfusion if their most recent platelet count is less than 20 x 109/L at the time of the planned procedure.
  Arms: Platelet
Other: 3- Platelet less than 30 x 109/L — Once randomized, the participant will receive a platelet transfusion if their most recent platelet count is less than 30 x 109/L at the time of the planned procedure.
  Arms: Platelet
Other: 4- Platelet less than 40 x 109/L — Once randomized, the participant will receive a platelet transfusion if their most recent platelet count is less than 40 x 109/L at the time of the planned procedure.
  Arms: Platelet
Other: 5- Platelet less than 50 x 109/L — Once randomized, the participant will receive a platelet transfusion if their most recent platelet count is less than 50 x 109/L at the time of the planned procedure.
  Arms: Platelet

SUMMARY:
The Canadian Critical Care Comparative Effectiveness Platform(e) d'Évaluation Clinique Comparée en soins Critiques (CEPEC) is an international multi-centered randomized adaptive platform clinical trial. CEPEC will evaluate supportive care interventions that are used routinely in intensive care units throughout the world.

DETAILED DESCRIPTION:
Many supportive therapies used daily in the ICU setting remain under-studied despite being resource-intensive. CEPEC aims to incorporate domains evaluating vasopressors, platelets, nutrition, sedation and analgesia, and other interventions.

VASOPRESSOR DOMAIN The investigators will investigate whether vasoactive medications should be used differently for different subgroups of patients who are in a state of cardiovascular shock (i.e. heterogeneity of treatment effects). Vasoactive medications are common in critically ill patients, and have considerable patient, hospital, and health system resource impact, but their use remains poorly supported by scientific evidence.

PLATELET DOMAIN Platelet transfusions are commonly prescribed to critically ill patients and have considerable patient, hospital, and health system resource impact, but remain poorly supported by scientific evidence. We propose to join a multicentre randomized clinical trial (T4P, ISRCTN79371664) addressing the optimal use of platelet transfusions for critically ill patients with thrombocytopenia in advance of invasive procedures. A multinational collaboration will ensure timely completion of this high-impact multicentre randomized clinical trial. The Canadian component of the T4P trial is embedded in the CEPEC platform as the Platelet Domain.

ELIGIBILITY:
VASOPRESSOR DOMAIN There is no minimum age limit in the Vasopressor Domain.

Inclusion criteria:

1. Ongoing vasopressor infusion to treat hypotension, or would be used to treat clinician-defined hypotension as part of usual care;
2. MAP <75 mmHg at any point (or lower than the upper value of the highest mean arterial pressure (MAP) target range activated locally);
3. Patient expected to be in the ICU for >48 hours.

Exclusion criteria:

1. Treating team does not have equipoise for at least two contiguous MAP target ranges in the CEPEC Vasopressor Domain;
2. Acute traumatic brain injury (within 7 days days or ongoing active treatment for elevated intracranial pressure);
3. Acute subarachnoid hemorrhage (within 21 days);
4. Acute spinal cord injury (within 7 days of injury or ongoing vasopressor therapy for suspected spinal cord ischemia);
5. Lung, heart, liver, kidney transplant recipient (within 7 days);
6. More than 24 hours since meeting inclusion criteria in the ICU;
7. Previously randomized into the CEPEC Vasopressor Domain or a confounding trial.

PLATELET DOMAIN

Inclusion criteria:

1. Adult patients (age ≥18 years) admitted to the ICU;
2. Latest platelet count in this hospital admission <50×109/L;
3. Planned to undergo a specified low-moderate bleeding risk invasive procedure.

Exclusion criteria:

1. Ongoing major hemorrhage requiring blood products and/or surgical/radiological intervention;
2. Intracranial hemorrhage within prior 72 hours;
3. Contraindications to platelet transfusion (e.g. thrombotic microangiopathies, heparin-induced thrombocytopenia, recent history of immune thrombocytopaenia, congenital platelet function defects);
4. Known advance decision of refusing blood/blood component transfusions;
5. Acute promyelocytic leukemia (APML);
6. Death perceived as imminent or admission for palliation;
7. Previously randomized into the CEPEC platelet domain or the T4P Trial;
8. Fulfilled all the inclusion criteria and none of the exclusion criteria ≥72 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6900 (Estimated)
Dates: Start 2025-03-23 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Vasopressor Domain - Composite endpoint | At hospital discharge up to day 30
  Incorporate mortality, persistent organ dysfunction (POD) in the intensive care unit (ICU), days in hospital, and disposition at hospital discharge.
Platelet Domain - All cause mortality | 90 days
  90-day all-cause mortality

SECONDARY OUTCOMES:
Vasopressor and Platelet Domains - Mortality | At hospital discharge up to day 30
Vasopressor and Platelet Domains - Persistent organ dysfunction (POD) in the ICU | At hospital discharge up to day 30
  POD is defined by the use of vasopressors, invasive mechanical ventilation, or new renal-replacement therapy whilst in ICU.
Vasopressor and Platelet Domains - Number of days without POD in the ICU | Up to day 30
  POD is defined by the use of vasopressors, invasive mechanical ventilation, or new renal-replacement therapy whilst in ICU.
Vasopressor and Platelet Domains - Disposition at hospital discharge | At hospital discharge up to day 30
  Increased level of care as indicated by change of address vs. return to baseline [previous home address]
Vasopressor and Platelet Domains - Number of days without POD in the ICU | At hospital discharge up to day 30
  POD is defined by the use of vasopressors, invasive mechanical ventilation, or new renal-replacement therapy whilst in ICU.
Platelet Domain - Mortality at discharge from hospital | Discharge from hospital
Platelet Domain - Mortality at 1 year | 1 year after randomization
Platelet Domain - Bleeding outcomes in hospital (major and fatal bleeds) | During hospitalization
Platelet Domain - Transfusion complications | During hospitalization
  Transfusion-associated circulatory overload, transfusion-related acute lung injury, infections, anaphylaxis
Platelet Domain - Days alive and at home at day 90 | 90 days
Platelet Domain - Number of days without persistent organ dysfunction in the ICU | Up to day 90
Platelet Domain - Health-related quality of life | 90 days
  Evaluated using EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Francois Lamontagne, MD, MSc, Principal Investigator — Université de Sherbrooke; Neill Adhikari, MDCM, MSc, Principal Investigator — Sunnybrook Research Institute
Locations (8):
- Canada (6):
  - Hamilton Health Sciences - Juravinski Hospital, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Scarborough Health Network, Scarborough Village, Ontario
  - Niagara Health, St. Catharines, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CIUSSS de l'Estrie - CHUS, Sherbrooke, Quebec
- Auckland City Hospital, Auckland, New Zealand
- Intensive Care National Audit and Research Centre (coordinating centre for sites in UK. Sites to be determined), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the CEPEC trial — https://cepec.ca/en